CLINICAL TRIAL: NCT05804903
Title: InvEstigation of the Safety and Performance of the NVT ALLEGRA Plus THV SysteM in Patients With Severe aortIc Stenosis or Failed suRgical Aortic bioprosthEsis
Brief Title: Investigation of the NVT ALLEGRA Plus THV System in Patients With Severe Aortic Stenosis or Failed Surgical Aortic Bioprosthesis
Acronym: EMPIRE-II
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NVT GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NVT06EMP2
Record Dates: First submitted 2023-03-14; First posted 2023-04-07 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Transcatheter Aortic Valve Implantation
Keywords: TAVI; Aortic valve stenosis; ALLEGRA Plus; IMPERIA; NVT
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAVI in severe calcified aortic stenosis or in failed surgical aortic bioprosthesis (Experimental)
  Interventions: Device: (ALLEGRA Plus Transcatheter Heart Valve) TAVI in severe calcified aortic stenosis or in failed surgical aortic bioprosthesis

INTERVENTIONS:
Device: (ALLEGRA Plus Transcatheter Heart Valve) TAVI in severe calcified aortic stenosis or in failed surgical aortic bioprosthesis — Implantation of the ALLEGRA Plus Transcatheter Heart Valve in severe calcified aortic stenosis or in failed surgical aortic bioprosthesis

SUMMARY:
The EMPIRE II study evaluates the safety and performance of the entire ALLEGRA THV System.

The primary safety endpoint is composite of all-cause mortality or stroke rates at 12 months. And the primary performance endpoint is device success at 7 days.

Based on the outcomes of a study with a similar device and considering a drop-out rate of 5%, 177 patients need to be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic severe calcific stenosis of a native aortic valve with an AVA ≤1.0 cm2 (or AVA index ≤0.6 cm2/m2), AND mean aortic pressure gradient ≥ 40mmHg OR maximal transaortic velocity ≥4.0m/s OR Doppler velocity index ≤0.25 on site-reported echocardiography OR symptomatic patients with degeneration of a surgical bioprosthetic valve (stenosis +/- insufficiency) on site-reported echocardiography
2. Local multi-disciplinary Heart Team and Central Screening Committee (CSC) agree on indication and eligibility for TAVI
3. Age ≥18 years
4. Patient has signed the Patient Informed Consent Form
5. Patient is willing and able to comply with requirements of the study, including all follow-up visits

Exclusion Criteria:

Patient will not be included if ANY one of the following conditions exists:

General:

1. Mean aortic annulus diameter as measured by pre-procedural CT or internal diameter of the bioprosthesis is <16.5 mm or >27 mm
2. Echocardiographic evidence of intracardiac thrombus or vegetation (site-reported)
3. Significant disease of the aorta that would preclude safe advancement of the ALLEGRA Plus THV System
4. Severe ilio-femoral vessel disease that would preclude safe placement of an 18 Fr introducer sheath or make endovascular access impossible
5. Porcelain aorta
6. Severe left ventricular dysfunction with ejection fraction (EF) <20% (site-reported)
7. Evidence of active endocarditis or other acute infections
8. Renal failure requiring continuous renal replacement therapy
9. Untreated clinically significant coronary artery disease requiring revascularization
10. Any percutaneous interventional procedure (e.g. PCI with stenting) within 14 days prior of the index procedure
11. Acute MI ≤30 days prior to the index procedure
12. Symptomatic carotid or vertebral artery disease requiring intervention or carotid/vertebral intervention within the preceding 45 days
13. Cerebrovascular accident (CVA) or transient ischemic attack (TIA) ≤6 months or prior CVA with moderate or severe disability (e.g. modified Rankin scale score >2)
14. History of bleeding diathesis or coagulopathy; acute blood dyscrasias as defined: thrombocytopenia (platelets <80,000/µl), acute anemia (hemoglobin <10 g/dl), leukopenia (WBC <3000/ µl)
15. Active peptic ulcer or gastrointestinal (GI) bleeding ≤3 months
16. Severe (greater than 3+) mitral insufficiency (site-reported)
17. Uncontrolled atrial fibrillation
18. Required emergency surgery for any reason
19. Known hypersensitivity to contrast media, which cannot be adequately pre-medicated or contraindication to anticoagulant or anti-platelet medication or to nitinol alloy or to bovine tissue
20. Life expectancy ≤12 months due to other medical illness
21. Currently participating in another investigational drug or device study
22. Hypertrophic obstructive cardiomyopathy
23. Pregnancy or intend to become pregnant during study participation

    Specific exclusions in patients with native aortic valve disease (site-reported):
24. Unicuspid or bicuspid aortic valve
25. Non-calcified aortic stenosis
26. Identified risk of coronary occlusion due to Sinus of Valsalva anatomy and/or bulky calcified aortic valve leaflets in close proximity to coronary ostia

    Specific exclusions in patients with degenerated surgical bioprosthetic aortic valves (valve-in-valve) (site-reported):
27. High risk of coronary occlusion
28. Partially detached leaflets that may obstruct a coronary ostium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Estimated)
Dates: Start 2023-11-24 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite of all-cause mortality or stroke rates | 12 months

SECONDARY OUTCOMES:
All-cause mortality rate | 7 days, 30 days, 6 months, 12 months, 2 years, 3 years , 4 years, 5 years
Cardiovascular mortality rate | 7 days, 30 days, 6 months, 12 months, 2 years, 3 years , 4 years, 5 years
Any stroke rate | 7 days, 30 days, 6 months, 12 months, 2 years, 3 years , 4 years, 5 years
Transient ischemic attack rate | 7 days, 30 days, 6 months, 12 months, 2 years, 3 years , 4 years, 5 years
Device success rate | 30 days
  Device success at 30 days (In-hospital may be used if 30-day data are not available):
  * Technical success
  * Freedom from mortality
  * Freedom from surgery or intervention related to the device (excluding permanent pacemaker) or to a major vascular or access-related or cardiac structural complication
  * Intended performance of the valve‡(mean gradient<20 mmHg, peakvelocity<3 m/s, Doppler velocity index ≥0.25, and less than moderate aortic regurgitation
Effective orifice area (EOA) as assessed by transthoracic echocardiogram (TTE) | 7 days, 30 days, 6 months, 12 months, 2 years, 3 years , 4 years, 5 years
  as determined by an independent Echo Core Lab
Transvalvular mean and peak pressure gradient as assessed by transthoracic echocardiogram (TTE) | 7 days, 30 days, 6 months, 12 months, 2 years, 3 years , 4 years, 5 years
  as determined by an independent Echo Core Lab
Transvalvular mean and peak pressure gradient as assessed by transthoracic | 7 days, 30 days, 6 months, 12 months, 2 years, 3 years , 4 years, 5 years
  as determined by an independent Echo Core Lab
NYHA classification | 7 days, 30 days, 6 months, 12 months, 2 years, 3 years , 4 years, 5 years
Life-threatening/major bleeding (BARC 3b or more) | 7 days, 30 days, 6 months, 12 months, 2 years, 3 years , 4 years, 5 years
Major vascular complications according to VARC-3 | 7 days, 30 days, 6 months, 12 months, 2 years, 3 years , 4 years, 5 years
Early safety profile according to VARC-3 | 30 days
Quality of life as assessed using the Kansas City Cardiomyopathy Questionnaire (KCCQ-12) | 7 days, 30 days, 6 months, 12 months, 2 years, 3 years , 4 years, 5 years
  Assessed with the Kansas City Cardiomyopathy Questionnaire (KCCQ-12). Patients are asked questions about physical limitation, symptom frequency, quality of life, and social limitation. Responses are given on a Likert scale that for each individual item is scored on a scale of 0-100 with higher scores indicating better health.
New pacemaker implantation rate | 7 days, 30 days, 6 months, 12 months, 2 years, 3 years , 4 years, 5 years

CONTACTS AND LOCATIONS:
Locations (7):
- Oulu University Hospital, Oulu, Finland
- Deutsches Herzzentrum Berlin, Berlin, State of Berlin, Germany
- Poland (2):
  - Klinika Kardiochirurgii, Gdansk
  - III Katedra Kardiologii, Katowice
- Spain (2):
  - Hospital La Paz, Madrid, Madrid
  - Reina Sofia Hospital, Córdoba
- Herzzentrum - Luzerner Kantonsspital, Lucerne, Switzerland